CLINICAL TRIAL: NCT04260308
Title: A Survey of Psychological Status of Medical Workers and Residents in the Context of 2019 Novel Coronavirus Pneumonia in Wuhan, China
Brief Title: A Survey of Psychological Status of Medical Workers and Residents in the Context of 2019 Novel Coronavirus Pneumonia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xianglin Yuan, professor, Huazhong University of Science and Technology
Other Study IDs: IRBID:TJ-C 20200107
Record Dates: First submitted 2020-02-03; First posted 2020-02-07 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Virus; Pneumonia
MeSH Terms: conditions — Pneumonia, Viral

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- residents: 1. Voluntary residents
  2. Can use mobile phone or computer
- medical staff: 1. Voluntary residents
  2. Can use mobile phone or computer

SUMMARY:
Due to the outbreak of 2019 Novel Coronavirus Pneumonia in Wuhan, Hubei province, medical staff and residents are facing great psychological pressure, the investigator plan to use electronic questionnaire to carry out investigation research.

DETAILED DESCRIPTION:
From December 2019, 12 cases of new coronavirus pneumonia broke out in Wuhan, and then the epidemic spread rapidly. Till February 1, 2020, there were 14446 confirmed cases in China, 19544 suspected cases, and 304 deaths. There were confirmed cases reported in 34 provincial administrative regions in China; 23 foreign countries reported new coronavirus pneumonia cases, 147 confirmed cases. In the face of the rapid spread of the epidemic, people's panic and anxiety have seriously affected the prevention and control of the epidemic. In the face of the occupational exposure risk and treatment brought by the sudden outbreak of the epidemic, the change of mental state of medical staff may affect the prevention and control of the epidemic. In order to help the epidemic prevention and control, the investigator plan to carry out investigation research.

ELIGIBILITY:
Inclusion Criteria:

* can use mobil phone or computer
* volunteer to take part in the investigation

Exclusion Criteria:

* can not use phone or computer
* unwilling to take part in the investigation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: medical staff and residents of China who is volunteer to take part in the investigation
Sampling Method: Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2020-02-03 (Actual); Primary Completion 2020-04-15 (Estimated); Study Completion 2020-04-20 (Estimated)

PRIMARY OUTCOMES:
GHQ-12(general health questionnaire-12) | 2 weeks
  GHQ-12(general health questionnaire-12): minimal score 0, maximal score 12, higher scores mean a better or worse outcome.

SECONDARY OUTCOMES:
IES-R(Impact of Event Scale-Revised) | 2 weeks
  IES-R(Impact of Event Scale-Revised):score range:0-88, the higher the worse

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital，Tongji Medical College Affiliated，Huazhong University of Science ＆ Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No